CLINICAL TRIAL: NCT03871855
Title: A Study of SHR-1702 Alone or With Camrelizumab in Participants With Advanced Relapsed/Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1702-I-101
Record Dates: First submitted 2019-02-17; First posted 2019-03-12 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A:SHR-1702 Dose Escalation (Experimental): SHR-1702 given intravenously (IV).
  Interventions: Drug: SHR-1702
- B:SHR-1702 Dose Expansion (Experimental): SHR-1702 given intravenously (IV).
  Interventions: Drug: SHR-1702
- C:SHR-1702 and Camrelizumab Dose Escalation (Experimental): SHR-1702 and Camrelizumab given intravenously (IV).
  Interventions: Drug: SHR-1702; Drug: Camrelizumab
- D:SHR-1702 and Camrelizumab Dose Expansion (Experimental): SHR-1702 and Camrelizumab given intravenously (IV).
  Interventions: Drug: SHR-1702; Drug: Camrelizumab

INTERVENTIONS:
Drug: SHR-1702 — Administered IV
Drug: Camrelizumab — Administered IV
  Arms: C:SHR-1702 and Camrelizumab Dose Escalation; D:SHR-1702 and Camrelizumab Dose Expansion

SUMMARY:
The purpose of this study is to evaluate the safety of SHR-1702 monotherapy or in combination with Camrelizumab among advanced solid tumor subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced relapsed/refractory solid tumors
* Must have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have an estimated life expectancy of 12 weeks, in judgement of the investigator；
* Must have at least 1 measurable lesion assessable using standard techniques by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Adequate hematologic and organ function
* Signed inform consent form

Exclusion Criteria:

* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Significant cardiovascular disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring
* History of autoimmune disease.
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid are permitted in the absence of active autoimmune disease.
* Positive test result for human immunodeficiency virus (HIV); Active hepatitis B or hepatitis C
* Active or untreated central nervous system (CNS) metastases
* Active infection within 2 weeks
* History of severe (or known) hypersensitivity to chimeric or humanized antibodies or fusion proteins
* Prior allogeneic bone marrow transplantation or solid organ transplant
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with DLTs | Approximately 28 Days

SECONDARY OUTCOMES:
ORR: Percentage of Participants With a CR or PR | Approximately 2 years
Safety and tolerability of SHR -1702 using Common Terminology Criteria for Adverse Events. | Dose Escalation Part -- Approximately 2 years
Immunogenicity as assessed by the presence of anti-drug antibodies | Approximately 2 years
Pharmacodynamic profile as assessed by receptor occupancy | Approximately 2 years
PK Parameter: Maximum Concentration (Cmax) | Approximately 2 years
PK Parameter: AUC, 0 to infinity | Approximately 2 years
PK Parameter: Clearance (CL) | Approximately 2 years
PK Parameter: Cmin at steady state (Cmin,ss) | Approximately 2 years
PK Parameter: Cmax at steady state (Cmax, ss) | Approximately 2 years
PK Parameter: terminal half-life (t1/2) | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China